CLINICAL TRIAL: NCT05495724
Title: An Open Label, Phase 2 Study of Disitamab Vedotin Combined With Tislelizumab for Patients With Her2 Overexpressing (IHC2+ or 3+) High-Risk Non-Muscle-Invasive Urothelial Bladder Carcinoma Which is Not Completely Resectable
Brief Title: Disitamab Vedotin Combined With Tislelizumab for Her2 Overexpressing High-Risk Non-Muscle-Invasive Urothelial Bladder Carcinoma Which is Not Completely Resectable
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRUCE-04
Record Dates: First submitted 2022-08-09; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Her2 Overexpressing High-Risk Non-Muscle Invasive Bladder Urothelial Carcinoma
Keywords: Disitamab Vedotin; Tislelizumab
MeSH Terms: interventions — disitamab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Disitamab Vedotin and Tislelizumab (Experimental): Disitamab Vedotin 120mg IV on day 1 in combination with Tislelizumab 200mg IV on day 2 every 3 weeks for 3 or 4 cycles followed by transurethral resection biopsy.
  Interventions: Drug: Disitamab Vedotin Tislelizumab
- Disitamab Vedotin (Other): Disitamab Vedotin 120mg IV on day 1 every 3 weeks for 3 or 4 cycles followed by transurethral resection biopsy.
  Interventions: Drug: Disitamab Vedotin

INTERVENTIONS:
Drug: Disitamab Vedotin Tislelizumab — Disitamab Vedotin 120mg will be administered on Day 1 of each cycle for 4 treatment cycles;Tislelizumab 200mg will be administered on Day 2 of each cycle for 4 treatment cycles.
  Other Names: KEYNOTE-057
  Arms: Disitamab Vedotin and Tislelizumab
Drug: Disitamab Vedotin — Disitamab Vedotin
  Arms: Disitamab Vedotin

SUMMARY:
This is a phase II study to determine the safety and efficacy of Disitamab Vedotin when given in combination with Tislelizumab as treatment for patients with Her2 overexpressing high-risk non-muscle-invasive bladder cancer (HR NMIBC) which is not completely resectable. Patients will receive treatment with Disitamab Vedotin in combination with tislelizumab every 3 weeks for 4 treatment cycles over 12 weeks followed by transurethral resection biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Urothelial carcinoma with Her2 IHC 2+ or 3+;
3. High-risk non-muscle-invasive urothelial carcinoma or high-risk non-muscle-invasive urothelial carcinoma as the main pathological component > 50%, difined as following:

   a. T1 b. High-grade Ta c.Carcinoma in situ(CIS);
4. Multi-point biopsy of bladder shows there are more than 2 section and over 3 points of pathological specimens are diagnosed as above, meanwhile, the tumor has to be diagnosed as not completely resectable by at least 2 senior urologist;
5. Agreed to provide tissue examination samples (for detection of PD-L1 expression, tumor mutation load, IHC, detection of DNA and RNA, etc;)
6. Organ function level must meet or under the support treatment meet the following requirements:

   * Hematological indexes: neutrophil count >= 1.5x10^9/L, platelet count >= 100x10^9/L, hemoglobin >= 9.0 g/dl;
   * Liver function: total bilirubin <=1.5 ULN, alanine aminotransferase and aspartate aminotransferase <=2.5 ULN（patient with metastatic liver cancer：aminotransferase <=5.0 ULN）;
   * Renal function: creatinine ≤ 1.5 times the upper limit of normal, and creatinine clearance ≥ 50 ml/min;
7. The subjects volunteered to join the study, signed informed consent, and had good compliance with follow-up;

Exclusion Criteria:

1. Active, known or suspected autoimmune diseases;
2. History of primary immunodeficiency;
3. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
4. Pregnant or lactating female patients;
5. Untreated acute or chronic active hepatitis B or hepatitis C infection. Under the condition of monitoring the virus copy number of patients receiving antiviral treatment, doctors can judge whether they are in line with the patients' individual conditions;
6. Prior use of immunosuppressive drugs within 4 weeks prior to the start of treatment, excluding nasal and inhaled corticosteroids or physiological doses of systemic steroids (i.e. not more than 10 mg / day prednisolone or other corticosteroids with the same physiological dose);
7. Known or suspected allergy to disitamab vedotin or tislelizumab;
8. Have a clear history of active tuberculosis;
9. Participating in other clinical researchers;
10. Men with reproductive capacity or women who are likely to become pregnant do not take reliable contraceptive measures;
11. Uncontrolled concurrent diseases, including but not limited to:

    * HIV infected (HIV antibody positive);
    * Severe infection in active stage or poorly controlled;
    * Evidence of serious or uncontrollable systemic diseases (such as severe mental, neurological, epilepsy or dementia, unstable or uncompensated respiratory, cardiovascular, liver or kidney diseases, uncontrolled hypertension [i.e. hypertension greater than or equal to CTCAE grade 2 after drug treatment]);
    * Patients with active bleeding or new thrombotic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2021-07-23 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) Rate | At the time of transurethral resection biopsy (within 9 or 12 weeks of the first dose of disitamab vedotin)

SECONDARY OUTCOMES:
Progress Free Survival（PFS） | up to 3 years
Recurrence Free Survival（RFS） | up to 3 years
Cystectomy-Free Survival (CFS) | up to 3 years
  defined from D1 of treatment until cystectomy
Duration of Response (DOR) | up to 3 years
Event-Free Survival（EFS） | up to 3 years
  defined from D1 of treatment until the time of any events，included progressive disease，discontinue treatment for any cause or death
Number of adverse events and severity by grade (CTCAE) | 12 weeks of treatment plus 30 days for toxicity followup
  Safety and toxicity will be characterized according to the reported adverse event (AE) profile using NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0, as well as a patient questionnaire derived from the Patient Reported Outcomes (PRO)-CTCAE and Patient Reported Outcomes Measurement Information System (PROMIS).
Her2 status | up to 3 years
PD-1 expression status | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Hailong Hu, Principal Investigator — Tianjin Medical University Second Hospital
Locations (1):
- Tianjin Medical University Second Hospital, Tianjin, Tianjin Municipality, China